CLINICAL TRIAL: NCT01444612
Title: Comparative Analysis of Injectable Anticoagulants for Thromboprophylaxis Post Cancer-related Surgery
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113164
Record Dates: First submitted 2011-06-23; First posted 2011-10-03 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Thrombosis, Venous
Keywords: cancer surgery; venous thromboembolism; hospitalization; anticoagulants; costs and cost analysis; thromboprophylaxis
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — Dalteparin; Enoxaparin; Fondaparinux; Heparin; calcium heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer-related surgery patient records: Healthcare claims records from patients aged 18 years or older with at least one primary inpatient discharge diagnosis of cancer and a cancer-related surgery during the hospitalization
  Interventions: Drug: dalteparin; Drug: enoxaparin; Drug: fondaparinux; Drug: unfractionated heparin

INTERVENTIONS:
Drug: dalteparin — An injectable anticoagulant medication for the prevention of VTE related to cancer surgery. Patients received dalteparin during one day prior to or two days after cancer-related surgery during the hospitalization.
  Other Names: Fragmin® is a registered trademark of Pfizer Health AB
Drug: enoxaparin — An injectable anticoagulant medication for the prevention of VTE related to cancer surgery. Patients received enoxaparin during one day prior to or two days after cancer-related surgery during the hospitalization.
  Other Names: Lovenox® is a registered trademark of Sanofi-Aventis
Drug: fondaparinux — An injectable anticoagulant medication for the prevention of VTE related to cancer surgery. Patients received fondaparinux during one day prior to or two days after cancer-related surgery during the hospitalization.
  Other Names: Arixtra® is a registered trademark of GlaxoSmithKline
Drug: unfractionated heparin — An injectable anticoagulant medication for the prevention of VTE related to cancer surgery. Patients unfractionated heparin received during one day prior to or two days after cancer-related surgery during the hospitalization.
  Other Names: heparin misc; heparin Ca; Calciparine; heparin beef lung; heparin Na; heparin/Ns; heparin/D5%; heparin/ns misc

SUMMARY:
Venous thromboembolism (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE), is a common post-operative complication. The effectiveness of fondaparinux compared with other injectable anticoagulants in VTE following major orthopedic and abdominal surgery has been evaluated in database studies; however, the effectiveness of injectable anticoagulant medications following cancer-related surgeries in the practice setting has not been as well documented.

The objective of this study is to analyze patient records from a national hospital database and compare the outcomes and costs between four types of injectable anticoagulant medications that were prescribed for the prevention of VTE following cancer-related surgery. This analysis will assess and quantify the outcomes, resource utilization, and cost of care for patients receiving fondaparinux, enoxaparin, dalteparin or unfractionated heparin. The outcomes of interest include the occurence of VTE, rates of major bleeds, medical resource utilization, and total costs (medical plus pharmacy).

The source of data for this study is the Premier Perspective Database™. This hospital claims database links de-identified inpatient medical, pharmacy, and billing data from more than 500 hospitals.

This study is a retrospective cohort study that uses propensity score matching to adjust for the differences between the numbers of patients treated with each medication.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* at least one record of a primary inpatient discharge diagnosis of cancer (index hospitalization)
* a procedure code for a cancer-related surgery during the index hospitalization
* a code for an anticoagulant treatment (dalteparin, enoxaparin, fondaparinux or unfractionated heparin (UFH)) as thromboprophylaxis therapy during the day prior to or two days after cancer-related surgery during the index hospitalization (this is the INDEX EVENT)

Exclusion Criteria:

* a record that the patient received more than one injectable anticoagulant on Day 1 of anticoagulant therapy
* a record that the patient received anticoagulant therapy prior to index anticoagulant
* a primary diagnosis code of DVT, PE, or major bleed
* evidence of an outpatient emergency department or hospital outpatient clinic visit that included a diagnosis code for DVT or PE during the 6 months prior to the index hospitalization
* patient records for patients transferred from another facility outside Premier system on index hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with at least one primary inpatient discharge diagnosis of cancer who experienced a cancer-related surgery during the hospitalization were the initial target population.
Sampling Method: Non-Probability Sample
Enrollment: 4068 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Rate of occurence of venous thromboembolism (VTE) during index hospitalization | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of hospital admission to the date of hospital discharge.
  VTE events were identified by International Classification of Disease-9 (ICD-9) codes for deep vein thrombosis (451.xx. 453.xx) and pulmonary embolism (415.xx) during the index hospitalization. Results will be calculated, reported as unadjusted, and adjusted to control for the effect of covariates on outcomes
Rate of occurence of major bleeding events during hospitalization | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of hospital admission to the date of hospital discharge.
  Major bleeding events were identified according to ICD-9 codes for major bleed (568.81, 430.xx, 431.xx, 432.xx, or 998.11) or other bleeding accompanied by more than 2 units of blood transfused (246.3, 286.5, 287.3, 287.4, 287.5, 287.8, 287.9, 459.0, 530.82, 569.3, 578.x, 596.7, 599.7, 719.1, 784.7, 784.8, 786.3, 958.2, or 997.02) as recorded in the billing file during the index hospitalization plus 1 month post discharge. Results will be calculated, reported as unadjusted, and adjusted to control for the effect of covariates on outcomes.
Rate of Hospital readmission rates | Data will be collected over a 5 year and 8 month period with this endpoint evaluated at one month following the date of hospital discharge
  Readmission rates were defined as a subsequent hospitalization for major bleeding or VTE that occurred within the follow-up period (discharge month plus 1 month).
Mean length of hospital stay in days | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of hospital admission to the date of hospital discharge.
  Length of hospital stay was obtained from the discharge record and was defined as the number of days from patient admission to the hospital for cancer-related surgery until discharge from the hospital.
Total cost of care for index hospitalization in United States (US) dollars | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of hospital admission to the date of hospital discharge.
  The mean total costs (medical plus pharmacy costs) from patient records in each antithrombotic cohort from the index hospitalization. Results will be calculated, reported as unadjusted, and adjusted to control for the effect of covariates on outcomes.

SECONDARY OUTCOMES:
Rate of occurence of VTE events during hospitalization plus 1 month post discharge. | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of admission for the index hospitalization to the end of the 1-month post-discharge follow-up period
  VTE events were identified according to ICD-9 codes for DVT and PE during the index hospitalization plus 1 month post discharge. Results will be calculated, reported as unadjusted, and adjusted to control for the effect of covariates on outcomes.
Rate of occurence of major bleeding events during hospitalization plus 1 month post discharge | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of admission for the index hospitalization to the end of the 1-month post-discharge follow-up period
  Major bleeding events were identified according to ICD-9 codes for hemoperitoneum bleed, intracranial hemorrhage/hemorrhagic stroke, hemorrhage complicating a procedure, or other bleeding accompanied by more than 2 units of blood transfused as recorded in the billing file during the index hospitalization plus 1 month post discharge. Results will be calculated, reported as unadjusted, and adjusted to control for the effect of covariates on outcomes.
Total cost of care for index hospitalization plus follow up in US dollars | Data will be collected over a 5 year and 8 month period with this endpoint evaluated from the date of the index hospitalization to the end of the 1-month post-discharge follow-up period
  The mean total costs (medical plus pharmacy costs) from patient records in each antithrombotic cohort from both the index hospitalization and the 1-month follow-up period. Results will be calculated, reported as unadjusted, and adjusted to control for the effect of covariates on outcomes

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline